CLINICAL TRIAL: NCT02534610
Title: Is There Any Analgesic Benefit From Preoperative vs. Postoperative Etoricoxib Administration in Total Knee Arthroplasty?
Brief Title: Analgesic Benefit of Preoperative vs. Postoperative Etoricoxib in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foisor Orthopedics Clinical Hospital (Other)
Responsible Party: Principal Investigator, Munteanu Ana Maria, MD, PhD, Medical Director, Foisor Orthopedics Clinical Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: AN010-13
Record Dates: First submitted 2015-08-20; First posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Postoperative Pain
Keywords: preemptive; postoperative pain; etoricoxib
MeSH Terms: conditions — Pain, Postoperative | interventions — Etoricoxib; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group ETORICOXIB PREOP (Experimental): Preoperative (1 h) per os (PO) 120 mg Etoricoxib (Arcoxia) and 1 placebo pill PO at the end of surgery.
  Interventions: Drug: Etoricoxib; Drug: Placebo
- Group ETORICOXIB POSTOP (Experimental): Preoperative (1 h) 1 placebo pill PO and 120 mg Etoricoxib PO at the end of surgery (Arcoxia).
  Interventions: Drug: Etoricoxib; Drug: Placebo
- Group PLACEBO (Placebo Comparator): 1 placebo pill PO 1 h preoperative and 1 placebo pill PO postoperative at the end of surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etoricoxib — 120 mg etoricoxib PO administered 1 h preoperative for group A; group B received 120 mg etoricoxib PO at the end of the surgery.
  Other Names: Arcoxia; Tauxib; Algix; Exxiv; Etozox
  Arms: Group ETORICOXIB POSTOP; Group ETORICOXIB PREOP
Drug: Placebo — Group A received 1 sham pill PO at the end of the surgery; group B received 1 sham pill PO 1 h preoperative and group C received sham pill PO 1 h preoperative and 1 sham pill PO at the end of the surgery.
  Other Names: Sham pill

SUMMARY:
Evaluation of the efficacy of preemptive versus postoperative administration of etoricoxib in total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
The investigators conducted a prospective randomized controlled study in 165 patients American Society of Anesthesiologists (ASA) score I-III scheduled for primary TKA, divided in 3 groups: group A (Etoricoxib 120 mg orally one hour before surgery), group B (Etoricoxib 120 mg orally at the end of surgery) and group C placebo. Surgery has been performed under spinal anesthesia.

All groups received postoperative analgesia when Numeric Rating Scale (NRS) over 3 with intravenous (IV) Perfalgan and morphine on demand for the following 48 h.

The effectiveness was evaluated by the time from the initiation of spinal anesthesia until the first analgesic dose at NRS > 3, the total amount of morphine in the first 24 and 48 hours postoperative, the side effects and necessary amount of adjuvant medication.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* weight (kilos) over 40 kg
* height (centimeters) over 155 cm
* non-anemic
* indication for primary TKA (total knee arthroplasty)

Exclusion Criteria:

* history of asthma
* peptic ulcer
* severe hepatic or renal dysfunction
* neuropathies
* bleeding disorders
* uncooperative
* drug abuse
* sensibility to etoricoxib
* paracetamol or morphine
* long acting nonsteroidal antiinflammatory drugs (NSAID) in the last 4 days preoperative
* cerebrovascular and peripheric vascular disease
* arterial hypertension (HTA) not adequately controlled
* congestive heart failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | At 48 hour postoperative
  Amount of IV and subcutaneous (SC) morphine (mg) required to reach NRS under 3

SECONDARY OUTCOMES:
Number of patients with side effects of drugs used | 48 hour postoperative
  number of patients with postoperative nausea and vomiting (PONV) or respiratory depression or gastric complaint or allergic reactions
Duration of analgesia | At 48 hours postoperative
  Time from spinal anesthesia until the first rescue morphine analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Munteanu Ana-Maria, MD, PhD, Principal Investigator — Foisor Orthopedics Clinical Hospital Bucharest; Stoica I Cristian, MD, Prof., Study Director — Foisor Orthopedics Clinical Hospital Bucharest
Locations (1):
- Foisor Orthopedics Clinical Hospital, Bucharest, Romania

REFERENCES:
- [Result] Buvanendran A, Kroin JS. Multimodal analgesia for controlling acute postoperative pain. Curr Opin Anaesthesiol. 2009 Oct;22(5):588-93. doi: 10.1097/ACO.0b013e328330373a. PMID 19606021
- [Result] Sinatra R. Role of COX-2 inhibitors in the evolution of acute pain management. J Pain Symptom Manage. 2002 Jul;24(1 Suppl):S18-27. doi: 10.1016/s0885-3924(02)00410-4. PMID 12204484
- [Result] Singer MA. Interaction of dibucaine and propranolol with phospholipid bilayer membranes-effect of alterations in fatty acyl composition. Biochem Pharmacol. 1977 Jan 1;26(1):51-7. doi: 10.1016/0006-2952(77)90129-0. No abstract available. PMID 188426
- [Result] Dahl JB, Moiniche S. Pre-emptive analgesia. Br Med Bull. 2004 Dec 13;71:13-27. doi: 10.1093/bmb/ldh030. Print 2004. PMID 15596866
- [Result] Moiniche S, Kehlet H, Dahl JB. A qualitative and quantitative systematic review of preemptive analgesia for postoperative pain relief: the role of timing of analgesia. Anesthesiology. 2002 Mar;96(3):725-41. doi: 10.1097/00000542-200203000-00032. No abstract available. PMID 11873051
- [Result] Lee BH, Park JO, Suk KS, Kim TH, Lee HM, Park MS, Lee SH, Park S, Lee JY, Ko SK, Moon SH. Pre-emptive and multi-modal perioperative pain management may improve quality of life in patients undergoing spinal surgery. Pain Physician. 2013 May-Jun;16(3):E217-26. PMID 23703420
- [Result] Derry S, Moore RA. Single dose oral celecoxib for acute postoperative pain in adults. Cochrane Database Syst Rev. 2013 Oct 22;2013(10):CD004233. doi: 10.1002/14651858.CD004233.pub4. PMID 24150982
- [Derived] Munteanu AM, Cionac Florescu S, Anastase DM, Stoica CI. Is there any analgesic benefit from preoperative vs. postoperative administration of etoricoxib in total knee arthroplasty under spinal anaesthesia?: A randomised double-blind placebo-controlled trial. Eur J Anaesthesiol. 2016 Nov;33(11):840-845. doi: 10.1097/EJA.0000000000000521. PMID 27454662